CLINICAL TRIAL: NCT07314554
Title: Recurrence Rate and Risk Factors After Endoscopic Resection of Gastric and Intestinal Polyps: A Retrospective and Prospective Cohort Study
Brief Title: Recurrence After Gastric and Intestinal Polyp Resection
Acronym: RAGIP
Status: Not yet recruiting | Type: Observational
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Zhaofeng Chen, Clinical Professor, LanZhou University
Other Study IDs: LDYYczf2025121801
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gastric Polyps; Intestinal Polyps; Colon Polyps; Colorectal Polyps; Adenomatous Polyps; Gastric Adenoma and Early Gastric Cancer; Colorectal Adenoma
Keywords: Polyp recurrence; Endoscopic resection; Polypectomy; Endoscopic mucosal resection; Endoscopic submucosal dissection; Risk factors; Surveillance; Follow-up; Adenoma; Gastric polyp; Colorectal polyp
MeSH Terms: conditions — Polyposis, Gastric; Intestinal Polyps; Colonic Polyps; Adenomatous Polyps; Stomach Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: Patients who underwent endoscopic polyp resection from January 2021 to December 2022, with retrospective data collection and follow-up through December 2025
- Prospective Cohort: Patients undergoing endoscopic polyp resection from October 2024 to December 2025, with prospective standardized data collection and follow-up through December 2028

SUMMARY:
This is a retrospective and prospective cohort study designed to evaluate the recurrence rate and identify risk factors after endoscopic resection of gastric and intestinal polyps.

BACKGROUND: Gastric and intestinal polyps are common digestive diseases with potential for malignant transformation. Although endoscopic resection is the standard treatment, recurrence rates range from 10-50%, and the mechanisms and risk factors remain unclear.

OBJECTIVES:

Primary: To assess short-term (1-year) and long-term (3-year) recurrence rates after endoscopic polyp resection Secondary: To identify independent risk factors and develop a recurrence risk prediction model

DESIGN: Mixed retrospective-prospective cohort study

* Retrospective cohort: Patients who underwent polyp resection from 2021-2022, with follow-up data through 2024
* Prospective cohort: Patients enrolled from 2024-2025, with standardized follow-up through 2028

SETTING: Single tertiary referral center with >10,000 endoscopic polyp resections performed since 2021

PARTICIPANTS: Approximately 1,600-1,800 adult patients (≥18 years) who underwent complete endoscopic resection of gastric or intestinal polyps

FOLLOW-UP:

* Short-term: 1 year post-resection (±2 months)
* Long-term: 3 years post-resection (±3 months)

MAIN OUTCOME: Recurrence rate defined as new polyp detection at original or different sites during endoscopic surveillance

POTENTIAL RISK FACTORS: Patient demographics, polyp characteristics (size, number, location, pathology), resection method, Helicobacter pylori status, lifestyle factors, and medication use

EXPECTED IMPACT: Results will inform personalized surveillance strategies and optimize resource allocation for post-polypectomy follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* First-time endoscopic examination (gastroscopy or colonoscopy) at the study center
* Pathologically confirmed polyp of any type (adenomatous, hyperplastic, inflammatory, fundic gland polyp, hamartomatous, serrated lesion)
* Complete endoscopic resection performed (including EMR, ESD, snare polypectomy, hot biopsy forceps, or argon plasma coagulation)
* Negative resection margins or complete resection assessed by pathology
* At least one follow-up endoscopic examination completed (for retrospective cohort) or willingness to complete follow-up (for prospective cohort)
* Complete baseline clinical data available

Exclusion Criteria:

* Hereditary polyposis syndromes (familial adenomatous polyposis, Lynch syndrome, Peutz-Jeghers syndrome, juvenile polyposis syndrome)
* Inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Previous history of gastric or colorectal cancer
* Cancer detected at initial resection (stage T1b or higher)
* Non-polyp pathology (e.g., submucosal tumors, normal mucosa)
* Incomplete resection with positive margins that were not re-treated
* Lost to follow-up with no available surveillance data (for retrospective cohort)
* Pregnancy at time of enrollment
* Inability or unwillingness to provide informed consent (for prospective cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (≥18 years) who underwent complete endoscopic resection of gastric or intestinal polyps at our tertiary referral center. This includes two cohorts: (1) Retrospective cohort: patients treated from 2021-2022 with existing follow-up data; (2) Prospective cohort: newly enrolled patients from 2024-2025. Eligible participants must have pathologically confirmed polyps (adenomatous, hyperplastic, inflammatory, fundic gland, serrated, or hamartomatous) with negative resection margins. The population represents a diverse group with varying polyp characteristics (size range: <5mm to >20mm; single or multiple polyps; gastric or colorectal locations) and different resection methods (EMR, ESD, snare polypectomy). Excluded are patients with hereditary polyposis syndromes, inflammatory bowel disease, prior gastrointestinal malignancy, or cancer detected at initial resection.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-02-25 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Short-term Recurrence Rate at 1 Year | 1 year post-resection (10-14 months acceptable)
  New polyp(s) detected by endoscopy and confirmed by pathology at 1-year follow-up. Includes both local recurrence (within 2cm of resection site) and metachronous polyps (>2cm from original site).
Long-term Recurrence Rate at 3 Years | 3 years post-resection (33-39 months acceptable)
  New polyp(s) detected by endoscopy and confirmed by pathology at 3-year follow-up. Includes both local recurrence and metachronous polyps.
Cumulative Recurrence Rate | Up to 3 years post-resection
  Overall recurrence rate combining 1-year and 3-year surveillance results

SECONDARY OUTCOMES:
Recurrence-free Survival Time | Up to 3 years
  Measured in months; censored at last follow-up for non-recurrent cases
Characteristics of Recurrent Polyps | At 1-year and 3-year follow-up
  Descriptive analysis of recurrent polyp features: Number, size, location, and pathological type of recurrent polyps.
Progression to High-grade Dysplasia or Cancer | Up to 3 years
  Pathologically confirmed progression: Proportion of participants developing high-grade dysplasia or invasive cancer during follow-up.
Re-treatment Rate | Up to 3 years
  Proportion of participants requiring repeat endoscopic or surgical treatment: Includes repeat polypectomy, endoscopic resection, or surgical resection
Identification of Independent Risk Factors | Analysis conducted after all follow-up completed (2029)
  Hazard ratios (HR) and 95% confidence intervals for each significant risk factor

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Lanzhou University, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sekiguchi M, Kakugawa Y, Matsumoto M, Matsuda T. A scoring model for predicting advanced colorectal neoplasia in a screened population of asymptomatic Japanese individuals. J Gastroenterol. 2018 Oct;53(10):1109-1119. doi: 10.1007/s00535-018-1433-7. Epub 2018 Jan 22. PMID 29359244
- [Background] Brenner H, Chang-Claude J, Jansen L, Knebel P, Stock C, Hoffmeister M. Reduced risk of colorectal cancer up to 10 years after screening, surveillance, or diagnostic colonoscopy. Gastroenterology. 2014 Mar;146(3):709-17. doi: 10.1053/j.gastro.2013.09.001. Epub 2013 Sep 5. PMID 24012982
- [Background] Click B, Pinsky PF, Hickey T, Doroudi M, Schoen RE. Association of Colonoscopy Adenoma Findings With Long-term Colorectal Cancer Incidence. JAMA. 2018 May 15;319(19):2021-2031. doi: 10.1001/jama.2018.5809. PMID 29800214
- [Background] Martinez ME, Baron JA, Lieberman DA, Schatzkin A, Lanza E, Winawer SJ, Zauber AG, Jiang R, Ahnen DJ, Bond JH, Church TR, Robertson DJ, Smith-Warner SA, Jacobs ET, Alberts DS, Greenberg ER. A pooled analysis of advanced colorectal neoplasia diagnoses after colonoscopic polypectomy. Gastroenterology. 2009 Mar;136(3):832-41. doi: 10.1053/j.gastro.2008.12.007. Epub 2008 Dec 9. PMID 19171141